CLINICAL TRIAL: NCT02269423
Title: A Phase 1 Randomized, Single-Center, Double-Blind, Placebo Controlled, Dose-Escalation Study to Evaluate the Safety and Immunogenicity of the BPSC-1001 (VSVΔG-ZEBOV) Ebola Virus Vaccine Candidate in Healthy Adult Subjects
Brief Title: Vaccine Treatment for Ebola Virus in Healthy Adults (V920-001)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Collaborators: BioProtection Systems Corporation (Industry); United States Department of Defense (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: V920-001; NLG0307 (WRAIR #2163) (Other: NewLink Genetics Corp.); V920-001 (Other: Merck Protocol Number)
Record Dates: First submitted 2014-10-10; First posted 2014-10-21 (Estimated); Results first posted 2019-10-23 (Actual); Last update posted 2019-10-23 (Actual); Status verified 2019-10

CONDITIONS: Ebola Virus

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- 3x10^6 plaque-forming units (pfu) Vaccine Cohort (Experimental): Participants will receive a 1-mL intramuscular injection of V920 3x10^6 pfu in one deltoid and a 1-mL intramuscular injection of placebo in the contralateral deltoid on Day 0.
  Interventions: Biological: V920; Other: Placebo
- 2x10^7 pfu Vaccine Cohort (Experimental): Participants will receive a 1-mL intramuscular injection of V920 2x10^7 pfu in one deltoid and a 1-mL intramuscular injection of placebo in the contralateral deltoid on Day 0.
  Interventions: Biological: V920; Other: Placebo
- 1x10^8 pfu Vaccine Cohort (Experimental): Participants will receive a 1-mL intramuscular injection of V920 1x10^8 pfu in one deltoid and a 1-mL intramuscular injection of placebo in the contralateral deltoid on Day 0.
  Interventions: Biological: V920; Other: Placebo
- Placebo Cohort (Placebo Comparator): Participants will receive a 1-mL intramuscular injection of placebo in each deltoid on Day 0.
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: V920 — Vesicular Stomatitis Virus (VSV)-based vaccine 1-mL injection containing 3x10^6, 2x10^7, or 1x10^8 pfu.
  Other Names: BPSC-1001
  Arms: 1x10^8 pfu Vaccine Cohort; 2x10^7 pfu Vaccine Cohort; 3x10^6 plaque-forming units (pfu) Vaccine Cohort
Other: Placebo — Normal saline placebo.

SUMMARY:
This is a study of the anti-Ebola vaccine vesicular stomatitis virus (VSV) ZEBOV (Zaire ebolavirus) also known as V920 and BPSC-1001. The purpose of this study is to test how safe the vaccine is in humans and how well it makes the human immune system cause an immune- or defense-response to Ebola virus. This vaccine will be studied at different doses.

DETAILED DESCRIPTION:
This study is being conducted to assess whether this vaccine is safe, and if it causes the body to create an infection-fighting response. Between 1994 and the present, there have been many Ebola virus outbreaks caused by 4 different strains of the virus, affecting mostly people living in central Africa and the health care providers trying to treat them. Ebola viruses are members of the filoviridae virus family, which also includes the dangerous Marburg virus. Ebola virus causes severe and often deadly infection called a viral hemorrhagic fever, characterized by organ failure, bleeding, and death.

To date, the virus is found primarily in Central and West Africa. It is not clear where these viruses come from, but it is thought that bats are the most likely source of the human outbreaks that occur. Once an outbreak occurs, the virus is spread from person to person through direct contact with infected blood or body fluids with an infected individual.

Given the recent increase in Ebola virus infections occurring in Africa, there is interest in making an effective vaccine to protect against the infection. V920/BPSC-1001 is an experimental Ebola vaccine candidate demonstrating protection against Ebola virus in animal experiments.

This is a Phase 1 study to evaluate a novel vaccine to Ebola using a live VSV replacing the gene encoding the G envelope glycoprotein with the gene encoding the envelope glycoprotein from the Zaire strain of Ebola (VSVΔG-ZEBOV also known as V920 and BPSC-1001). This phase 1 protocol provides a first-in-human study to evaluate the safety and toxicity of V920/BPSC-1001 in healthy adult participants. Participants will be randomized to receive V920/BPSC-1001 or Placebo by intramuscular injection. Three dose levels will be assessed with follow-up visits through 180 days after the injection.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adult male or non-pregnant, non-lactating female, ages 18 to 50 (inclusive) at the time of screening
* Have provided written informed consent before screening
* Free of clinically significant health problems, as determined by pertinent medical history and clinical examination prior to entry into the study
* Available, able, and willing to participate for all study visits and procedures
* Males and females who are willing to practice abstinence from sexual intercourse, or willing to use effective methods of contraception, from at least 30 days prior to vaccination until study end.
* Be willing to minimize blood and body fluid exposure of others for 7 days after vaccination
* Score at least 80% on the Comprehension Assessment test

Exclusion Criteria:

* History of prior infection with a filovirus or prior participation in a filovirus vaccine trial
* History of prior infection with VSV or receipt of a VSV vectored vaccine
* Is a healthcare worker who has direct contact with patients
* Has a house-hold contact (HHC) who is immunodeficient, Human Immunodeficiency Virus (HIV)-positive, pregnant, has an unstable medical condition, or is under the age of 5 years
* Is a childcare worker who has direct contact with children 5 years of age or younger
* Directly prepares food in the food industry
* History of employment in an industry involved in contact with ruminant animals, veterinary sciences, or other potential exposure to VSV
* Planned or frequent contact with animals at-risk of VSV infection (e.g. cattle, horses, pigs, mules, etc.)
* History of employment or activity which involves potential contact with filoviruses
* History of severe local or systemic reactions to any vaccination or a history of severe allergic reactions
* Known allergy to the components of the BPSC1001 vaccine product
* Receipt of investigational product up to 30 days prior to enrollment or ongoing participation in another clinical trial
* Receipt of licensed vaccines within 30 days of planned study immunization
* Ongoing participation in another clinical trial
* Ability to observe possible local reactions at the eligible injections sites (deltoid region) is, in the opinion of the investigator, unacceptably obscured due to a physical condition or permanent body art
* Acute or chronic, clinically significant psychiatric, hematologic, pulmonary, cardiovascular, or hepatic or renal functional abnormality as determined by the investigator based on medical history, physical exam, electrocardiogram, and/or laboratory screening test. This would include a known hemoglobinopathy or coagulation abnormality.
* Any baseline laboratory screening tests which is outside of acceptable range as defined in the protocol.: alanine aminotransferase, aspartate aminotransferase, creatinine, hemoglobin, platelet count, total white blood cell count, urine protein, urine occult blood, urine glucose
* Any serologic evidence of hepatitis B or C infection
* Any confirmed or suspected immunosuppressive or immunodeficient condition, including HIV infection, cytotoxic therapy in the previous 5 years, and/or diabetes
* Any chronic or active neurologic disorder, including migraines, seizures, and epilepsy, excluding a single febrile seizure as a child
* Have an active malignancy or history of metastatic or hematologic malignancy
* Suspected or known alcohol and/or illicit drug abuse within the past 5 years
* Moderate or severe illness and/or fever >100.4F within one week prior to vaccination
* Pregnant or lactating female, or female who intends to become pregnant during the study period
* Administration of immunoglobulins and/or any blood products within the 120 days preceding study entry or planned administration during the study period
* History of blood donation within 60 days of enrollment or plans to donate within the study period
* Administration of chronic (defined as more than 14 days) immunosuppressants or other immune modifying drugs within 6 months of study entry. (For corticosteroids, this will mean prednisone, or equivalent, greater than or equal to 0.5 mg/kg/day, Intranasal and topical steroids are allowed)
* Unwilling to allow storage and use of blood for future vaccine research
* Any other significant finding that in the opinion of the investigator would increase the risk of the individual having an adverse outcome from participating in this study

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 39 (Actual)
Dates: Start 2014-10-13 (Actual); Primary Completion 2015-08-25 (Actual); Study Completion 2015-08-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Derived] Coller BG, Blue J, Das R, Dubey S, Finelli L, Gupta S, Helmond F, Grant-Klein RJ, Liu K, Simon J, Troth S, VanRheenen S, Waterbury J, Wivel A, Wolf J, Heppner DG, Kemp T, Nichols R, Monath TP. Clinical development of a recombinant Ebola vaccine in the midst of an unprecedented epidemic. Vaccine. 2017 Aug 16;35(35 Pt A):4465-4469. doi: 10.1016/j.vaccine.2017.05.097. Epub 2017 Jun 21. PMID 28647166
- [Derived] Regules JA, Beigel JH, Paolino KM, Voell J, Castellano AR, Hu Z, Munoz P, Moon JE, Ruck RC, Bennett JW, Twomey PS, Gutierrez RL, Remich SA, Hack HR, Wisniewski ML, Josleyn MD, Kwilas SA, Van Deusen N, Mbaya OT, Zhou Y, Stanley DA, Jing W, Smith KS, Shi M, Ledgerwood JE, Graham BS, Sullivan NJ, Jagodzinski LL, Peel SA, Alimonti JB, Hooper JW, Silvera PM, Martin BK, Monath TP, Ramsey WJ, Link CJ, Lane HC, Michael NL, Davey RT Jr, Thomas SJ; rVSVDeltaG-ZEBOV-GP Study Group. A Recombinant Vesicular Stomatitis Virus Ebola Vaccine. N Engl J Med. 2017 Jan 26;376(4):330-341. doi: 10.1056/NEJMoa1414216. Epub 2015 Apr 1. PMID 25830322

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | 3x10^6 Plaque-forming Units (Pfu) Vaccine Cohort | 2x10^7 Pfu Vaccine Cohort | 1x10^8 Pfu Vaccine Cohort | Placebo Cohort
Started | 10 | 10 | 10 | 9
Completed | 10 | 9 | 10 | 8
Not Completed | 0 | 1 | 0 | 1
Not completed — Discontinued due to change in residence | 0 | 1 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 3x10^6 Plaque-forming Units (Pfu) Vaccine Cohort | 2x10^7 Pfu Vaccine Cohort | 1x10^8 Pfu Vaccine Cohort | Placebo Cohort | Total
Number analyzed (Participants) | 10 | 10 | 10 | 9 | 39
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 10 | 10 | 10 | 9 | 39
  >=65 years | 0 | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 3 | 2 | 4 | 12
  Male | 7 | 7 | 8 | 5 | 27
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 1 | 0 | 3
  Not Hispanic or Latino | 9 | 9 | 9 | 9 | 36
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 2 | 0 | 0 | 1 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 3 | 5 | 5 | 3 | 16
  White | 4 | 5 | 5 | 5 | 19
  More than one race | 1 | 0 | 0 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With One or More Solicited Local Treatment-Emergent Adverse Events (TEAE)
Description: An adverse event (AE) is defined as any untoward medical occurrence in a participant which does not necessarily have a causal relationship with study vaccine. A treatment-emergent adverse event (TEAE) is defined as an AE that starts or worsens on or after the date and time of the study vaccination. Local reactogenicity signs and symptoms include pain, erythema (redness), and induration (swelling). The number of participants that experienced at least one solicited local TEAE was assessed. Solicited TEAEs occurred from the time of each injection through 14 days following the procedure, facilitated with the use of a memory aid to record participant observations.
Time Frame: Up to 14 days postvaccination
Population: All randomized participants who received study vaccination (V920 dose level or placebo).
Measure: Count of Participants; unit: Participants
Arm/Group | 3x10^6 Plaque-forming Units (Pfu) Vaccine Cohort | 2x10^7 Pfu Vaccine Cohort | 1x10^8 Pfu Vaccine Cohort | Placebo Cohort
Number analyzed (Participants) | 10 | 10 | 10 | 9
Participants | 8 | 8 | 10 | 3

2. Primary Outcome: Number of Participants With One or More Solicited Local Treatment-Emergent Adverse Events (TEAE) by Severity
Description: An AE is defined as any untoward medical occurrence in a participant which does not necessarily have a causal relationship with study vaccine. A TEAE is defined as an AE that starts or worsens on or after the date and time of the study vaccination. Local reactogenicity signs and symptoms include pain, erythema (redness), and induration (swelling). AEs were assessed for severity by the investigator according to a toxicity grading scale based on the FDA's Guidance for Industry "Toxicity Grading Scale for Healthy Adult and Adolescent Volunteers Enrolled in Preventive Vaccine Clinical Trials": Grade 1=Mild; Grade 2=Moderate; Grade 3=Severe; Grade 4=Potentially life-threatening. The number of participants that experienced at least one solicited local TEAE was summarized by grade. Solicited TEAEs occurred from the time of each injection through 14 days following the procedure, facilitated with the use of a memory aid to record participant observations.
Time Frame: Up to 14 days postvaccination
Population: All randomized participants who received study vaccination (V920 dose level or placebo).
Measure: Count of Participants; unit: Participants
Arm/Group | 3x10^6 Plaque-forming Units (Pfu) Vaccine Cohort | 2x10^7 Pfu Vaccine Cohort | 1x10^8 Pfu Vaccine Cohort | Placebo Cohort
Number analyzed (Participants) | 10 | 10 | 10 | 9
Participants
  Grade 1 (Mild) | 6 | 7 | 9 | 3
  Grade 2 (Moderate) | 2 | 1 | 1 | 0
  Grade 3 (Severe) | 0 | 0 | 0 | 0
  Grade 4 (Potentially life-threatening) | 0 | 0 | 0 | 0

3. Primary Outcome: Number of Participants With One or More Solicited Systemic Treatment-Emergent Adverse Events (TEAE)
Description: An adverse event (AE) is defined as any untoward medical occurrence in a participant which does not necessarily have a causal relationship with study vaccine. A treatment-emergent adverse event is defined as an AE that starts or worsens on or after the date and time of the study vaccination. Systemic reactogenicity signs and symptoms include pyrexia (subjective and objective fever), chills, hyperhidrosis (sweats), myalgia, arthralgia, fatigue, headache, and gastrointestinal symptoms including nausea, vomiting, abdominal pain, and/or diarrhea. The number of participants that experienced at least one solicited systemic TEAE was assessed. Solicited TEAEs occurred from the time of each injection through 14 days following the procedure, facilitated with the use of a memory aid to record participant observations.
Time Frame: Up to 14 days postvaccination
Population: All randomized participants who received study vaccination (V920 dose level or placebo).
Measure: Count of Participants; unit: Participants
Arm/Group | 3x10^6 Plaque-forming Units (Pfu) Vaccine Cohort | 2x10^7 Pfu Vaccine Cohort | 1x10^8 Pfu Vaccine Cohort | Placebo Cohort
Number analyzed (Participants) | 10 | 10 | 10 | 9
Participants | 9 | 7 | 9 | 6

4. Primary Outcome: Number of Participants With One or More Solicited Systemic Treatment-Emergent Adverse Events (TEAE) by Severity
Description: An AE is defined as any untoward medical occurrence in a participant which does not necessarily have a causal relationship with study vaccine. A TEAE is defined as an AE that starts or worsens on or after the date and time of the study vaccination. Systemic reactogenicity signs and symptoms include pyrexia (subjective and objective fever), chills, hyperhidrosis (sweats), myalgia, arthralgia, fatigue, headache, and gastrointestinal symptoms including nausea, vomiting, abdominal pain, and/or diarrhea. AEs were assessed for severity by the investigator as follows: Grade 1=Mild; Grade 2=Moderate; Grade 3=Severe; Grade 4=Potentially life-threatening. The number of participants that experienced at least 1 solicited systemic TEAE was summarized by grade. Solicited TEAEs occurred from the time of each injection through 14 days following the procedure, facilitated with the use of a memory aid to record participant observations.
Time Frame: Up to 14 days postvaccination
Population: All randomized participants who received study vaccination (V920 dose level or placebo).
Measure: Count of Participants; unit: Participants
Arm/Group | 3x10^6 Plaque-forming Units (Pfu) Vaccine Cohort | 2x10^7 Pfu Vaccine Cohort | 1x10^8 Pfu Vaccine Cohort | Placebo Cohort
Number analyzed (Participants) | 10 | 10 | 10 | 9
Participants
  Grade 1 (Mild) | 3 | 2 | 2 | 5
  Grade 2 (Moderate) | 3 | 3 | 4 | 1
  Grade 3 (Severe) | 3 | 2 | 3 | 0
  Grade 4 (Potentially life-threatening) | 0 | 0 | 0 | 0

5. Primary Outcome: Number of Participants With One or More Unsolicited Treatment-Emergent Adverse Events (TEAE)
Description: An adverse event (AE) is defined as any untoward medical occurrence in a participant which does not necessarily have a causal relationship with study vaccine. A treatment-emergent adverse event is defined as an AE that starts or worsens on or after the date and time of the study vaccination. The number of participants that experienced at least one unsolicited TEAE was assessed. Unsolicited AEs occurred from the time of injection through 28 days following injection.
Time Frame: Up to 28 days postvaccination
Population: All randomized participants who received study vaccination (V920 dose level or placebo).
Measure: Count of Participants; unit: Participants
Arm/Group | 3x10^6 Plaque-forming Units (Pfu) Vaccine Cohort | 2x10^7 Pfu Vaccine Cohort | 1x10^8 Pfu Vaccine Cohort | Placebo Cohort
Number analyzed (Participants) | 10 | 10 | 10 | 9
Participants | 10 | 9 | 9 | 8

6. Primary Outcome: Number of Participants With One or More Vaccination-Related Unsolicited Treatment-Emergent Adverse Events (TEAE)
Description: An adverse event (AE) is defined as any untoward medical occurrence in a participant which does not necessarily have a causal relationship with study vaccine. A treatment-emergent adverse event is defined as an AE that starts or worsens on or after the date and time of the study vaccination. A related TEAE is defined as a TEAE that was possibly, probably, or definitely related to the vaccination as assessed by the investigator. The number of participants that experienced at least one unsolicited TEAE related to study vaccination was assessed.
Time Frame: Up to 28 days postvaccination
Population: All randomized participants who received study vaccination (V920 dose or placebo).
Measure: Count of Participants; unit: Participants
Arm/Group | 3x10^6 Plaque-forming Units (Pfu) Vaccine Cohort | 2x10^7 Pfu Vaccine Cohort | 1x10^8 Pfu Vaccine Cohort | Placebo Cohort
Number analyzed (Participants) | 10 | 10 | 10 | 9
Participants | 8 | 8 | 7 | 6

7. Primary Outcome: Number of Participants With One or More Vaccination-Related Unsolicited Treatment-Emergent Adverse Events (TEAE) by Severity
Description: An adverse event (AE) is defined as any untoward medical occurrence in a participant which does not necessarily have a causal relationship with study vaccine. A treatment-emergent adverse event is defined as an AE that starts or worsens on or after the date and time of the study vaccination. A related TEAE is defined as a TEAE that was possibly, probably, or definitely related to the vaccination as assessed by the investigator. AEs were assessed for severity by the investigator according to a toxicity grading scale based on the FDA's Guidance for Industry "Toxicity Grading Scale for Healthy Adult and Adolescent Volunteers Enrolled in Preventive Vaccine Clinical Trials": Grade 1=Mild; Grade 2=Moderate; Grade 3=Severe; Grade 4=Potentially life-threatening. The number of participants that experienced at least one unsolicited TEAE related to study vaccination was summarized by grade.
Time Frame: Up to 28 days postvaccination
Population: All randomized participants who received study vaccination (V920 dose level or placebo).
Measure: Count of Participants; unit: Participants
Arm/Group | 3x10^6 Plaque-forming Units (Pfu) Vaccine Cohort | 2x10^7 Pfu Vaccine Cohort | 1x10^8 Pfu Vaccine Cohort | Placebo Cohort
Number analyzed (Participants) | 10 | 10 | 10 | 9
Participants
  Grade 1 (Mild) | 1 | 2 | 2 | 5
  Grade 2 (Moderate) | 3 | 3 | 3 | 1
  Grade 3 (Severe) | 4 | 3 | 2 | 0
  Grade 4 (Potentially life-threatening) | 0 | 0 | 0 | 0

8. Primary Outcome: Number of Participants With Early Study Discontinuation Due to an Adverse Event
Description: An adverse event (AE) is defined as any untoward medical occurrence in a participant which does not necessarily have a causal relationship with study vaccine. The number of participants prematurely withdrawing from the study due to an AE was assessed.
Time Frame: Up to 28 days postvaccination
Population: All randomized participants who received study vaccination (V920 dose level or placebo).
Measure: Count of Participants; unit: Participants
Arm/Group | 3x10^6 Plaque-forming Units (Pfu) Vaccine Cohort | 2x10^7 Pfu Vaccine Cohort | 1x10^8 Pfu Vaccine Cohort | Placebo Cohort
Number analyzed (Participants) | 10 | 10 | 10 | 9
Participants | 0 | 0 | 0 | 0

9. Secondary Outcome: Geometric Mean Titers of ZEBOV Envelope Glycoprotein-specific Binding Antibodies
Description: The Geometric Mean Titers (GMT) of ZEBOV-specific Immunoglobulin G antibodies were measured by unqualified ZEBOV immunoglobulin (IgG) enzyme-linked immunosorbent assay (ELISA). For titers expressed in ELISA Units/mL, the lower level of quantitation (LLOQ) was 58.84. ZEBOV IgG titers at baseline (Day 0) and analysis Days 7, 14, 28, 56, 84, and 180 were summarized by V920 vaccine dose level and placebo as the mean of log10 titers, transformed into GMT. The geometric standard deviation (GSD) for the GMT at each visit was obtained by exponentiating the standard deviation for the mean of log (base 10) transformed titers.
Time Frame: Baseline, Days 7, 14, 28, 56, 84 and 180 post-vaccination
Population: All randomized participants who were vaccinated and had an evaluable Day 28 immunogenicity result following vaccination and who did not have any protocol deviations that influenced interpretation of immunogenicity endpoints for the specified measurement and timeframe.
Measure: Geometric Mean (Standard Deviation); unit: ELISA Units/mL
Arm/Group | 3x10^6 Plaque-forming Units (Pfu) Vaccine Cohort | 2x10^7 Pfu Vaccine Cohort | 1x10^8 Pfu Vaccine Cohort | Placebo Cohort
Number analyzed (Participants) | 10 | 10 | 10 | 9
ELISA Units/mL
  Baseline (Day 0) | 29.42 (1.00) | 29.42 (1.00) | 33.85 (1.56) | 35.09 (1.70)
  Day 7 | 29.42 (1.00) | 29.42 (1.00) | 29.42 (1.00) | 34.92 (1.67)
  Day 14: number analyzed (Participants) | 10 | 10 | 9 | 9
  Day 14 | 225.23 (2.15) | 360.14 (4.04) | 621.68 (5.45) | 35.24 (1.72)
  Day 28 | 911.79 (2.09) | 1570.84 (2.40) | 2662.23 (2.88) | 36.54 (1.92)
  Day 56: number analyzed (Participants) | 10 | 9 | 10 | 9
  Day 56 | 1425.16 (2.14) | 2031.53 (2.02) | 2677.04 (3.59) | 31.81 (1.26)
  Day 84: number analyzed (Participants) | 10 | 9 | 10 | 9
  Day 84 | 1245.40 (1.96) | 1816.81 (2.14) | 2374.33 (4.36) | 31.85 (1.27)
  Day 180: number analyzed (Participants) | 10 | 9 | 10 | 7
  Day 180 | 1494.69 (3.21) | 1177.40 (2.22) | 1658.50 (3.13) | 39.44 (2.17)
Statistical Analysis 1: Comparison: 3x10^6 Plaque-forming Units (Pfu) Vaccine Cohort vs Placebo Cohort; Day 28; Test type: Other; p < 0.001, ANOVA — p-values are pairwise comparisons of log-transformed titers between each V920 dose, between each V920 dose and placebo, between all V920 dose levels combined and placebo and are from an ANOVA model; Adjustments for multiple comparisons were not performed
Statistical Analysis 2: Comparison: 2x10^7 Pfu Vaccine Cohort vs Placebo Cohort; Day 28; Test type: Other; p < 0.001, ANOVA — [p-value comment as in outcome 9, analysis 1]; Adjustments for multiple comparisons were not performed
Statistical Analysis 3: Comparison: 1x10^8 Pfu Vaccine Cohort vs Placebo Cohort; Day 28; Test type: Other; p < 0.001, ANOVA — [p-value comment as in outcome 9, analysis 1]; Adjustments for multiple comparisons were not performed
Statistical Analysis 4: Comparison: 3x10^6 Plaque-forming Units (Pfu) Vaccine Cohort vs 2x10^7 Pfu Vaccine Cohort; Day 28; Test type: Other; p = 0.161, ANOVA — [p-value comment as in outcome 9, analysis 1]; Adjustments for multiple comparisons were not performed
Statistical Analysis 5: Comparison: 3x10^6 Plaque-forming Units (Pfu) Vaccine Cohort vs 1x10^8 Pfu Vaccine Cohort; Day 28; Test type: Other; p = 0.008, ANOVA — [p-value comment as in outcome 9, analysis 1]; Adjustments for multiple comparisons were not performed
Statistical Analysis 6: Comparison: 2x10^7 Pfu Vaccine Cohort vs 1x10^8 Pfu Vaccine Cohort; Day 28; Test type: Other; p = 0.173, ANOVA — [p-value comment as in outcome 9, analysis 1]; Adjustments for multiple comparisons were not performed

10. Secondary Outcome: Geometric Mean Titers of ZEBOV-specific Neutralizing Antibodies
Description: The Geometric Mean Titers (GMT) of ZEBOV-specific neutralizing antibodies were measured by pseudovirion neutralization assays (PsVNA). Titers were reported for PsVNA50 values which were derived from the reciprocal of the dilution that resulted in a 50% decrease in luciferase activity. The LLOQ for the PsVNA was 20. If the PsVNA was reported ≤20, the numeric portion of the titer was divided by 2 for statistical purposes, which could result in a reported GMT <20.0. PsVNA50 titers at baseline (Day 0) and analysis Days 7, 14, 28, 56, and 180 were summarized by V920 vaccine dose level and placebo as the mean of log10 titers, transformed into GMT. The geometric standard deviation (GSD) for the GMT at each visit was obtained by exponentiating the standard deviation for the mean of log (base 10) transformed titers.
Time Frame: Baseline, Days 7, 14, 28, 56, and 180 post-vaccination
Population: as for outcome 9
Measure: Geometric Mean (Standard Deviation); unit: titer
Arm/Group | 3x10^6 Plaque-forming Units (Pfu) Vaccine Cohort | 2x10^7 Pfu Vaccine Cohort | 1x10^8 Pfu Vaccine Cohort | Placebo Cohort
Number analyzed (Participants) | 10 | 10 | 10 | 9
titer
  Baseline | 10.0 (1.00) | 10.0 (1.00) | 10.0 (1.00) | 10.0 (1.00)
  Day 7 | 10.0 (1.00) | 10.0 (1.00) | 10.0 (1.00) | 10.0 (1.00)
  Day 14: number analyzed (Participants) | 10 | 10 | 9 | 9
  Day 14 | 46.0 (2.83) | 216.5 (3.29) | 140.4 (3.58) | 10.0 (1.00)
  Day 28 | 222.8 (3.20) | 468.0 (3.96) | 447.0 (2.10) | 10.0 (1.00)
  Day 56: number analyzed (Participants) | 10 | 9 | 10 | 9
  Day 56 | 137.7 (2.38) | 170.3 (1.86) | 218.6 (3.06) | 10.0 (1.00)
  Day 180: number analyzed (Participants) | 9 | 9 | 10 | 8
  Day 180 | 29.1 (4.23) | 23.0 (2.90) | 46.2 (3.06) | 10.0 (1.00)
Statistical Analysis 1: Comparison: 3x10^6 Plaque-forming Units (Pfu) Vaccine Cohort vs Placebo Cohort; Day 28; Test type: Other; p < 0.001, ANOVA — [p-value comment as in outcome 9, analysis 1]; Adjustments for multiple comparisons were not performed
Statistical Analysis 2: Comparison: 2x10^7 Pfu Vaccine Cohort vs Placebo Cohort; Day 28; Test type: Other; p < 0.001, ANOVA — [p-value comment as in outcome 9, analysis 1]; Adjustments for multiple comparisons were not performed
Statistical Analysis 3: Comparison: 1x10^8 Pfu Vaccine Cohort vs Placebo Cohort; Day 28; Test type: Other; p < 0.001, ANOVA — [p-value comment as in outcome 9, analysis 1]; Adjustments for multiple comparisons were not performed
Statistical Analysis 4: Comparison: 3x10^6 Plaque-forming Units (Pfu) Vaccine Cohort vs 2x10^7 Pfu Vaccine Cohort; Day 28; Test type: Other; p = 0.102, ANOVA — [p-value comment as in outcome 9, analysis 1]; Adjustments for multiple comparisons were not performed
Statistical Analysis 5: Comparison: 3x10^6 Plaque-forming Units (Pfu) Vaccine Cohort vs 1x10^8 Pfu Vaccine Cohort; Day 28; Test type: Other; p = 0.124, ANOVA — [p-value comment as in outcome 9, analysis 1]; Adjustments for multiple comparisons were not performed
Statistical Analysis 6: Comparison: 2x10^7 Pfu Vaccine Cohort vs 1x10^8 Pfu Vaccine Cohort; Day 28; Test type: Other; p = 0.918, ANOVA — [p-value comment as in outcome 9, analysis 1]; Adjustments for multiple comparisons were not performed

11. Secondary Outcome: Number of Participants With Vaccine Viremia
Description: The number of participants with viremia detected by recombinant vesicular stomatitis virus (rVSV) reverse transcription polymerase chain reaction (PCR) of blood specimens was assessed.
Time Frame: Days 1, 3, 7, and 14 post-vaccination
Population: All randomized subjects who were vaccinated and had an evaluable Day 28 immunogenicity result following vaccination and who did not have any protocol deviations that influenced interpretation of immunogenicity endpoints.
Measure: Count of Participants; unit: Participants
Arm/Group | 3x10^6 Plaque-forming Units (Pfu) Vaccine Cohort | 2x10^7 Pfu Vaccine Cohort | 1x10^8 Pfu Vaccine Cohort | Placebo Cohort
Number analyzed (Participants) | 10 | 10 | 10 | 9
Participants
  Day 1 | 10 | 10 | 10 | 0
  Day 3 | 10 | 10 | 9 | 1
  Day 7 | 1 | 2 | 3 | 0.0
  Day 14 | 0.0 | 0.0 | 0.0 | 0.0

12. Secondary Outcome: Number of Participants With Vaccine Shedding/Excretion in Saliva or Urine
Description: The number of participants with viremia detected by rVSV reverse transcription PCR of saliva or urine specimens was assessed.
Time Frame: Days 1, 3, 7, and 14 post-vaccination
Population: as for outcome 11
Measure: Count of Participants; unit: Participants
Arm/Group | 3x10^6 Plaque-forming Units (Pfu) Vaccine Cohort | 2x10^7 Pfu Vaccine Cohort | 1x10^8 Pfu Vaccine Cohort | Placebo Cohort
Number analyzed (Participants) | 10 | 10 | 10 | 9
Participants
  Day 1 | 0 | 0 | 1 | 0
  Day 3 | 1 | 0 | 0 | 0
  Day 7 | 1 | 1 | 0 | 0
  Day 14 | 0 | 1 | 0 | 0

13. Primary Outcome: Number of Participants With One or More Serious Adverse Event
Description: An adverse event is defined as any untoward medical occurrence in a participant which does not necessarily have a causal relationship with study vaccine. A serious adverse event (SAE) is an AE that results in death, is life-threatening, results in a persistent or significant disability or incapacity, results in or prolongs an existing hospitalization, is a congenital anomaly or birth defect, or is another important medical event. The number of participants that experienced one or more SAE was summarized.
Time Frame: Up to 180 days postvaccination
Population: All participants who received study vaccination (V920 dose level or placebo).
Measure: Count of Participants; unit: Participants
Arm/Group | 3x10^6 Plaque-forming Units (Pfu) Vaccine Cohort | 2x10^7 Pfu Vaccine Cohort | 1x10^8 Pfu Vaccine Cohort | Placebo Cohort
Number analyzed (Participants) | 10 | 10 | 10 | 9
Participants | 0 | 0 | 0 | 0

14. Secondary Outcome: Mean Copy Number of Vector RNA (Vector Viremia)
Description: Although the protocol specified a secondary endpoint that included the mean copy number of vector RNA (vector viremia), the Polymerase Chain Reaction (PCR) test used for the study reported a qualitative rather than a quantitative outcome, so the proportion of participants with viremia is reported instead of the mean copy number of vector RNA. Qualitative results are therefore reported in Outcome Measures 12 and 13.
Time Frame: Up to 14 days postvaccination
Population: Although the plan specified in the protocol was to describe vector viremia by summarizing simple mean copy numbers of vector RNA, this data was not collected as the PCR results were qualitative rather than quantitative and were assessed in outcome measures # 12 and #13 instead.
Arm/Group | 3x10^6 Plaque-forming Units (Pfu) Vaccine Cohort | 2x10^7 Pfu Vaccine Cohort | 1x10^8 Pfu Vaccine Cohort | Placebo Cohort
Number analyzed (Participants) | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Up to 180 days
Description: All participants that received study vaccination (V920 dose or placebo) and had safety follow-up data.
  The AEs in this section are combined (solicited and unsolicited) events. The results reported under the Outcome Measures are based on specific conditions (separated for solicited and unsolicited AEs and days postvaccination). For example, the terms "pyrexia" and "hyperhidrosis" in this section correspond to "objective fever, "subjective fever", and "sweats" as reported in the Outcome Measures.
Arm/Group | 3x10^6 Plaque-forming Units (Pfu) Vaccine Cohort | 2x10^7 Pfu Vaccine Cohort | 1x10^8 Pfu Vaccine Cohort | Placebo Cohort
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/10 | 0/10 | 0/9
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10 | 0/10 | 0/9
Other Adverse Events (participants affected / at risk) | 10/10 | 10/10 | 10/10 | 9/9
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 3x10^6 Plaque-forming Units (Pfu) Vaccine Cohort (N=10) | 2x10^7 Pfu Vaccine Cohort (N=10) | 1x10^8 Pfu Vaccine Cohort (N=10) | Placebo Cohort (N=9)
Anemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lymphopenia (Blood and lymphatic system disorders) | 7 (7) | 0 (0) | 2 (2) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Blepharospasm (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Photophobia (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 2 (2) | 2 (2) | 2 (3) | 1 (2)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 2 (2) | 1 (1)
Nausea (Gastrointestinal disorders) | 2 (2) | 3 (4) | 2 (3) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Chills (General disorders) | 3 (3) | 4 (4) | 7 (7) | 1 (1)
Fatigue (General disorders) | 6 (9) | 4 (5) | 7 (12) | 4 (4)
Injection site bruising (General disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Injection site pain (General disorders) | 8 (8) | 8 (11) | 10 (15) | 4 (5)
Injection site swelling (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 4 (7) | 4 (6) | 8 (13) | 1 (1)
Pharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pharyngitis streptococcal (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sinusitis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 2 (2) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Blood urea increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hemoglobin decreased (Investigations) | 0 (0) | 0 (0) | 3 (3) | 2 (2)
Lymphocyte count decreased (Investigations) | 0 (0) | 7 (7) | 5 (5) | 0 (0)
Platelet count decreased (Investigations) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Prothrombin time prolonged (Investigations) | 1 (1) | 1 (1) | 1 (1) | 3 (3)
White blood cell count decreased (Investigations) | 2 (2) | 2 (2) | 3 (3) | 1 (1)
White blood cell count increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Neutrophil count decreased (Investigations) | 1 (1) | 2 (2) | 3 (3) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 5 (6) | 2 (2)
Myalgia (Musculoskeletal and connective tissue disorders) | 6 (6) | 4 (4) | 6 (6) | 1 (1)
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dizziness postural (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 6 (11) | 6 (8) | 8 (14) | 7 (10)
Sinus headache (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Phobia (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hematuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Proteinuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nasal dryness (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rhinorrhea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 4 (4) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
All data may be published in the open medical or military literature with the identity of the subjects protected. Anyone desiring to publish or present data obtained during the conduct of the study will conform to WRAIR, USAMRIID, and the sponsor's policies and then forward the publication for review to the sponsor and usarmy.detrick.medcom-usamrmc.list.clearances@mail.mil prior to submission.